CLINICAL TRIAL: NCT03674853
Title: Clinical Study of Wuling Capsule in the Treatment of Chronic Tinnitus With Emotional Disorder
Brief Title: The Study of Wuling Capsule in Treatment Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20172099-1
Record Dates: First submitted 2018-09-13; First posted 2018-09-18 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-05

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — wuling; ginaton; gamma-oryzanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wuling Capsule group (Experimental): Patients who were treated with Wuling Caspule
  Interventions: Drug: Wuling Capsule
- Oryzanol group (Active Comparator): Patients who were treated with oryzanol
  Interventions: Drug: Oryzanol

INTERVENTIONS:
Drug: Wuling Capsule — take Wuling Capsule in experiment group for 2 months
  Other Names: Ginaton
  Arms: Wuling Capsule group
Drug: Oryzanol — take oryzanol in active comparator group for 2 months
  Other Names: Ginaton
  Arms: Oryzanol group

SUMMARY:
To evaluate the effect of psychological/mental factors on the severity of subjective tinnitus, to observe the efficacy and safety of Wuling capsule in the treatment of chronic subjective tinnitus with emotional disorders, and to evaluate the control rate of tinnitus complications, such as depression, anxiety and insomnia, and the improvement of patients'quality of life.

DETAILED DESCRIPTION:
To evaluate the effect of psychological/mental factors on the severity of subjective tinnitus, to observe the efficacy and safety of Wuling capsule in the treatment of chronic subjective tinnitus with emotional disorders, and to evaluate the control rate of tinnitus complications, such as depression, anxiety and insomnia, and the improvement of patients'quality of life. Patients with chronic tinnitus complicated with mild to moderate anxiety or depression were randomly divided into two groups. The experimental group was given oral treatment with Wuling capsule, and the control group was given gurusu treatment. The improvement of tinnitus, sleep, anxiety and depression in patients was evaluated at 2,4 and 8 weeks after treatment, respectively, and the efficacy of Wuling capsule in improving tinnitus combined with anxiety, depression and tinnitus was analyzed。

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus with a history longer than 6 months;
* 7 < HAMD score < 24 and / or 7 < HAMA score < 21;
* No antianxiety, depression or antipsychotic treatment within 2 weeks.

Exclusion Criteria:

* objective tinnitus;
* tinnitus with defined causes;
* accompanied with acute infection, acute trauma, perioperative, chronic disease in the acute stage;
* with mental illness family history;
* HAMD score greater than 24 points or HAMA score greater than 21 points;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
the change of severity of tinnitus | 8 weeks
  tinnitus handicap index is to evaluate the severity of tinnitus

SECONDARY OUTCOMES:
the change of anxiety level | 8 weeks
  Hamilton anxiety scale is to evaluate the anxiety level
the change of depression level | 8 weeks
  Hamilton depression scale is to evaluate the depression level

CONTACTS AND LOCATIONS:
Overall Officials: Zha Dingjun, doctor, Study Chair — First Affiliated Hospital of Fourth Military Medical University
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No